CLINICAL TRIAL: NCT04753372
Title: Effectiveness and Safety of Low Dose Rivaroxaban Plus Aspirin in Patients With Chronic Coronary Syndrome and High Ischemic Risk
Brief Title: Rivaroxaban Plus Aspirin in Patients With Chronic Coronary Syndrome and High Ischemic Risk
Status: Completed | Type: Observational
Sponsor: Maatschap Cardiologie Zwolle (Other)
Collaborators: Diagram B.V. (Other)
Responsible Party: Sponsor
Other Study IDs: Dutch Rivaroxaban CCS Registry
Record Dates: First submitted 2020-12-22; First posted 2021-02-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease (CAD); Peripheral Arterial Disease (PAD)
Keywords: Coronary Artery Disease (CAD); peripheral arterial disease (PAD); high ischemic risk
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rivaroxaban 2.5 MG [Xarelto] — rivaroxaban 2.5mg bid on top of ASA for CAD and/or PAD
  Other Names: acetylsalicylic acid (ASA)

SUMMARY:
Registry to describe the impact in terms of effectiveness and safety of the combination treatment of rivaroxaban 2.5 mg twice daily with aspirin on clinical outcomes and practices in a real-life Dutch patient population that are at high risk of ischemic events.

DETAILED DESCRIPTION:
This study is a national multicentre (~15 sites), prospective, single-arm, observational study in patients treated with rivaroxaban 2.5mg bid on top of ASA75-100mg OD (N=1000). Female and male patients with a diagnosis of CCS and/or symptomatic PAD will be enrolled in the (outpatient) clinic after the decision for treatment with rivaroxaban 2.5mg bid, co-administered with acetylsalicylic acid has been made by the treating physician.

The primary effectiveness endpoint is a composite of:

* Major Adverse Cardiac Events (MACE including stroke, cardiovascular mortality and myocardial infarction)
* Clinically driven coronary, peripheral or carotid revascularization
* Stent thrombosis at one year

The primary safety endpoint is Major Bleeding at one year. These major bleeding complications are analysed according to the International Society on Thrombosis and Haemostasis (ISTH) criteria as a composite of fatal bleeding, symptomatic bleeding into a critical organ (such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome), bleeding causing a fall in haemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.

The secondary endpoints will be:

* Occurrence (and date) of stroke
* Occurrence (and date) of myocardial infarction
* Occurrence (and date) of cardiovascular death
* Occurrence (and date) of coronary revascularization procedures (PCI, CABG).
* Occurrence (and date) of peripheral revascularization procedures.
* Occurrence (and date) of carotid revascularization procedures.
* Occurrence (and date) of minor bleeding complications (according to ISTH)

In addition, all bleeding events including minor bleedings according to ISTH definitions will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patient.
* Diagnosis of CAD and/or PAD and high risk of ischemic events.

  * Patients at high risk of ischaemic events include the following:
  * CAD + PAD
  * CAD + Recurrent MI (Previous MI followed by second MI)
  * CAD + diabetes mellitus (all types)
  * CAD + chronic kidney disease with eGFR 30-59 ml/min/1.73 m2 (CKD-EPI formula)
  * CAD + heart failure (ejection fraction ≥30% - 50%) and New York Heart Association (NYHA) class I or II;)
  * CAD + CHA2DS2VaSc ≥ 3 (for men) or ≥ 4 (for women)
* Patients can only be enrolled in the study if the decision to treat with rivaroxaban plus ASA has been made by the treating physician in advance and independent of study inclusion, however within 4 weeks prior to study inclusion.
* Treatment according to local marketing authorization, with rivaroxaban 2.5 mg [BID] and 80mg ASA / 100mg Carbasalate calcium. Treatment of rivaroxaban started within 4 weeks prior or 4 weeks after study inclusion.
* Patients who are willing to participate in this study (signed informed consent).

Exclusion Criteria:

* Hypersensitivity/allergy and known contraindication to ASA/Carbasalate calcium or rivaroxaban
* Patients with recent major bleeding, active bleeding, or history with:

  * History of major clinical bleeding or known coagulopathy
  * History of intracerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke
  * Known severe liver dysfunction
* Patients that have received any organ transplant or await any organ transplant
* Patient with anemia (Hb < 6.0 mmol/L)
* Patient with active malignancy
* Patients with ejection fraction < 30% and/or New York Heart Association (NYHA) class III or IV
* Patients with eGFR < 30 ml/min/1.73m2 or undergoing dialysis
* Patients with liver failure accompanied with coagulopathy ( incl. Child-Pugh B and C)
* Patients with concomitant use of other anticoagulants or antiplatelet drugs
* Pregnant or lactating female
* Patients currently participating in another investigational drug or drug-coated device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients with a diagnosis of CCS and/or symptomatic PAD will be enrolled in the (outpatient) clinic within 4 weeks after the decision for treatment with rivaroxaban 2x2.5mg plus ASA (75-100mg) has been made by the investigator (according to label (indicated for the prevention of atherothrombotic events in adult patients with coronary artery disease (CAD) or symptomatic peripheral artery disease (PAD) at high risk of ischemic events)) and who consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures | one year
  The primary efficacy endpoint is a composite of 1) Major Adverse Cardiovascular Events (MACE), which is a composite endpoint of cardiovascular mortality, myocardial infarction and stroke, 2) clinically driven coronary, peripheral or carotid revascularization, and 3) stent thrombosis, that will be reported at 1 year.
  The primary safety endpoint is major bleeding according to the International Society on Thrombosis and Haemostatsis (ISTH) criteria that will be reported at 1 year. It is a composite of 1) fatal bleeding, 2) symptomatic bleeding into a critical organ (such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome), 3) bleeding causing a fall in haemoglobin level of 2 g/dL (1.24 mmol/L) or more, or 4) leading to transfusion of two or more units of whole blood or red cells.

SECONDARY OUTCOMES:
Secondary Outcome Measures | one year
  The secondary efficacy and safety endpoint is the incidence of individual endpoints, that will be reported at 1 year:
  1. Occurrence (and date) of stroke
  2. Occurrence (and date) of myocardial infarction
  3. Occurrence (and date) of cardiovascular death
  4. Occurrence (and date) of coronary revascularization procedures (PCI, CABG).
  5. Occurrence (and date) of peripheral revascularization procedures.
  6. Occurrence (and date) of carotid revascularization procedures.
  7. Occurrence (and date) of minor bleeding complications (according to ISTH)

CONTACTS AND LOCATIONS:
Overall Officials: Rik Hermanides, MD, PhD, Principal Investigator — Isala
Locations (12):
- Netherlands (12):
  - Jeroen Bosch hospital, 's-Hertogenbosch
  - OLVG, Amsterdam
  - Rijnstate hospital, Arnhem
  - Medisch Spectrum Twente, Enschede
  - Zuyderland Medical Center, Heerlen
  - Isala Klinieken, location Meppel, Meppel
  - St. Antonius hospital, Nieuwegein
  - Haaglanden Medisch Centrum, The Hague
  - Hagaziekenhuis, The Hague
  - Elisabeth-Tweesteden hospital, Tilburg
  - VieCuri, Venlo
  - Isala hospital, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided